CLINICAL TRIAL: NCT01615770
Title: Behavioral Maintenance Treatment for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joel D Killen, Principle Investigator, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: SU-09282010-6951; R01DA017441 (NIH)
Record Dates: First submitted 2010-10-07; First posted 2012-06-11 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open Label CBT and Pharmacotherapy (No Intervention): All study participants received 8 weeks of cognitive and behavioral cessation and relapse prevention skills training (CBT) and nicotine patch therapy combined with 9 weeks of bupropion SR therapy. Following open-label, this group received general supportive therapy delivered via four telephone calls made to participants over a 12-week period.
- Behavioral: cognitive behavior therapy (Experimental): All study participants received 8 weeks of cognitive and behavioral cessation and relapse prevention skills training (CBT) and nicotine patch therapy combined with 9 weeks of bupropion SR therapy. Following open-label treatment, half the participants received an additional 12 weeks of CBT that combined clinic-based skills training sessions, voicemail monitoring and telephone counseling
  Interventions: Behavioral: cognitive behavior therapy

INTERVENTIONS:
Behavioral: cognitive behavior therapy — At each clinic session, staff met with participants individually for 30 minutes to develop cognitive and behavioral skills to resist urges to smoke. Staff used self-efficacy questionnaires to assess participants' confidence in their abilities to resist urges to smoke in specific situations and behavioral worksheets to help participants articulate treatment plans to be used in managing their behavior in these situations without smoking. Those participants randomized to extended CBT continued to work with treatment staff individually on the development and use of cognitive and behavioral cessation and relapse prevention skills. Treatment sessions, lasting approximately 30 minutes, were conducted at the San Jose clinic site at weeks 8, 12, 16 and 20.
  Arms: Behavioral: cognitive behavior therapy

SUMMARY:
Our primary goal is to examine the effectiveness of a multi-factor maintenance treatment strategy in promoting longer-term smoking abstinence. The investigators will also conduct secondary analyses of mediators and moderators of treatment response.

DETAILED DESCRIPTION:
400 adult smokers will be randomized. Our primary goal is to examine the effectiveness of a multi-factor maintenance treatment strategy in promoting longer-term smoking abstinence. All smokers will receive the same "Acute Phase Treatment" that combines nicotine patch, bupropion and intensive self-regulatory skills training. Nicotine patches will be provided for 8 weeks and bupropion and skills training will be provided for of 9 weeks. Participants will then enter a "Maintenance Treatment Phase" during which half (n=200) will receive three individualized relapse prevention training sessions spread over a 12 week period. They will also receive 12 weeks of self-administered RPT administered via written treatment modules. Finally, telephone counseling will be provided in conjunction with an Interactive Voice Response system (IVR) that will allow early detection of smoking "slips" and rapid response by treatment staff. The other half (n=200) will be assigned to a control condition that consists of three counselor-led sessions of "supportive therapy" spread over a 12 week period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult cigarette smokers smoking at least 10 cigarettes per day

Exclusion Criteria:

* Currently pregnant
* Currently breastfeeding
* Currently diagnosed with a seizure disorder, major depression, liver disease, kidney disease, congestive heart failure
* History of a seizure, seizure disorder, significant head trauma or central nervous system tumor
* Family history of seizures
* Currently using intravenous drugs
* Currently using any drugs (marijuana, alcohol, cocaine, opiates, stimulants, etc.) on a daily basis
* Currently using any over-the-counter stimulants and anorectics (diet pills)
* Currently on bupropion (Wellbutrin, Wellbutrin SR) or other antidepressants, monoamine oxidase inhibitors, antipsychotics, benzodiazepines, theophylline, systemic steroids or levodopa
* Currently on NRT or bupropion (Zyban)
* Current or past diagnosis of anorexia nervosa or bulimia nervosa
* Previous allergic response to bupropion or NRT
* Previous failed quit attempt using NRT and bupropion in combination

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2004-02; Primary Completion 2006-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
expired-air carbon monoxide confirmed 7-day point prevalence smoking abstinence | 52 weeks
  expired-air carbon monoxide < 10 ppm and self report of no smoking for 7 consecutive days prior to assessment

SECONDARY OUTCOMES:
depression symptoms | 52 weeks
  symptoms of depression measured with the CES-D

CONTACTS AND LOCATIONS:
Overall Officials: Joel D Killen, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford Stop Smoking Program, San Jose, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey SR, Hammer SA, Bryson SW, Schatzberg AF, Killen JD. Using treatment process data to predict maintained smoking abstinence. Am J Health Behav. 2010 Nov-Dec;34(6):801-10. doi: 10.5993/ajhb.34.6.14. PMID 20604703
- [Result] Killen JD, Fortmann SP, Schatzberg AF, Arredondo C, Murphy G, Hayward C, Celio M, Cromp D, Fong D, Pandurangi M. Extended cognitive behavior therapy for cigarette smoking cessation. Addiction. 2008 Aug;103(8):1381-90. doi: 10.1111/j.1360-0443.2008.02273.x. PMID 18855829